CLINICAL TRIAL: NCT06207630
Title: Prevention of the Risk of Complete Sternotomy Scar Dehiscence in Cardiac Surgery: A Randomized, Open-label Multicenter Clinical Investigation Comparing Negative Pressure Wound Therapy (NPWT) vs. Standard Dressing
Brief Title: Prevention of the Risk of Complete Sternotomy Scar Dehiscence in Cardiac Surgery: A Clinical Investigation Comparing Negative Pressure Wound Therapy (NPWT) vs. Standard Dressing
Acronym: PRISTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRISTER
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Complete Vertical Midline Sternotomy / Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard dressing group (Active Comparator): Use dry dressing, made with sterile compresses, then a glued dressing
  Interventions: Device: Dressing Device
- NPWT 3/7d dressing group (Experimental): Use of a PICO® dressing
  Interventions: Device: Dressing Device
- NPWT 7d dressing group (Experimental): Use of a PREVENA® dressing
  Interventions: Device: Dressing Device

INTERVENTIONS:
Device: Dressing Device — Use of a dress at the end of surgery in the operating room, making sure not to stick it on the openings of the chest drains.

SUMMARY:
Mediastinitis is the most feared infectious complication after cardiac surgery. Several risk factors are known such as: obesity, diabetes, chronic obstructive pulmonary disease, double breast sampling, immunodeficiency, corticosteroid therapy, reoperation, chest radiotherapy, and dialysis. Three modes of contamination are described: intraoperative contamination, hematogenous dissemination during sepsis, gradual contamination from cutaneous dehiscence. It is important and simple to fight against this third mode. The dehiscence of the sternotomy scar represents a gateway and facilitates bacterial colonization and is a risk factor for infection of the surgical site. These skin disunities lead to an increase in health care costs due to extension of hospital stay, the cost of repeated nursing care, surgical revision, and the need for increased follow-up. They delay cardiac rehabilitation and return home. It is estimated that these simple disunities occur in more than 15% of cases, although fortunately they rarely result in mediastinitis. While the use of NPWT for the prevention of wound healing complications is permitted, its benefit has not been demonstrated. Its action is multiple with a reduction in the rate of repair of dressings and therefore of soiling, drainage of the wound, limitation of maceration, acceleration of healing. The use of NPWT as a dressing for sternotomies could prevent skin breakdown, and therefore superficial and deep surgical site infections.

Two types of NPWT devices exist, corresponding to 2 different types of treatment: the 7-day NPWT without dressing repair but with reservoir (PREVENA®), the NPWT with 3-day repair without reservoir (PICO®).

Given the cost and widespread use of NPWT for chirurgical site infection prophylaxis, it is important to conduct randomized trials to assess the expected benefit of these NPWTs designed for use on clean, closed surgical incisions. In cardiac surgery, its benefit has only been shown in a high-risk population: surgery for Coronary Artery Bypass Graft (CABG).

The present clinical investigation will be the first randomized, multicenter trial comparing the efficacy and safety of NPWT versus standard dressing in preventing the risk of scar dehiscence after cardiac surgery, in a standard population.

The patients will be followed for 90 days (3 months).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing scheduled or semi-urgent cardiac surgery, with or without extracorporeal circulation.
* Patients managed by complete vertical median sternotomy.
* Patients benefiting from a Social Security scheme or benefiting from it through a third party.
* Informed consent signed by the patient after clear and complete information about the clinical investigation.

All patients included in this clinical investigation must not have any of the non-inclusion criteria listed below:

Exclusion Criteria:

* Known allergy to one of the dressings: PREVENA®, PICO® or standard dressing
* Patient with a contraindication to PICO® dressing
* Patient with a contraindication to PREVENA® dressing:

  * Sensitivity to silver
* Patient with a history of cardiac surgery prior to inclusion
* Patient with skin infection (folliculitis) of the sternotomy site before the operation.
* Urgency and extreme urgency (patient operated within 24 hours of admission).
* Patient already participating in a clinical investigation whose main objective or secondary objectives are likely to have an impact on the main objective of this clinical investigation
* Patient with antibiotherapy ongoing (endocarditis patients)
* Minimal sternotomy (8-10 cm)
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy), or having a positive pregnancy test at inclusion
* The inability of the patient to complete informed consent before any study procedure
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Complete median sternotomy wound cutaneous dehiscence | 30 postoperative days
  Complete median sternotomy wound cutaneous dehiscence in cardiac surgery during the first 30 postoperative days will be assessed by tablet calibrated photos analyzed by an independent blinded staff.

SECONDARY OUTCOMES:
The number of dressing repairs | Between 7 and 90 postoperative days
The length of initial hospital stay | Between 7 and 90 postoperative days
The occurrence of an infection of the surgical site and its classification | At Day 90
The use of an anti-infectious treatment and its duration. | Between 7 and 90 postoperative days
The incidence of postoperative mediastinitis defined by dehiscence of the sternum with positive sternal samples. | At Day 90
The incidence of surgical revision for dehiscence of the surgical wound at D90. | At Day 90
  Collection of all operations involving surgical revision of the sternotomy wound.
The number of rehospitalizations (including consultations), and their duration. | At Day 90
The nurse's satisfaction with the use of the 3 types of dressing during dressing repair by means of a standardized questionnaire. | 7 postoperative days
  The nurse's satisfaction with the use of the 3 types of dressing during dressing repair by means of a standardized questionnaire consisting in four questions rated from 1 (not satisfied) to 5 (totally satisfied): Are you satisfied with application of this dressing? Are you satisfied with management of the surgical wound? Are you satisfied with follow-up on the wound? Are you satisfied with the visual appearance of the surgical wound?
The surgeon's satisfaction with the wound by means of a standardized questionnaire. | 7 postoperative days
  The surgeon's satisfaction with the wound by means of a standardized questionnaire consisting in four questions rated from 1 (not satisfied) to 5 (totally satisfied): Are you satisfied with application of this dressing? Are you satisfied with management of the surgical wound? Are you satisfied with follow-up on the wound? Are you satisfied with the visual appearance of the surgical wound? .
The incremental cost-utility ratio expressed in costs per quality-adjusted life-year (QALY) gained. | Between 7 and 90 postoperative days
  Medico-economic assessment will be assessed by evaluation of hospital and extra-hospital costs (number of days in hospital, consultations, re-hospitalisations, imaging, biology and drugs), dressing costs and patient quality of life by EQ-5D-5L. The proposed analysis will be a cost-utility analysis because health-related quality of life is a significant outcome of the studied interventions.
The incremental cost-effectiveness ratio expressed in costs per post-operative complication avoided | Between 7 and 90 postoperative days
  Resource utilization data will be collected prospectively for all patients enrolled in the clinical investigation. The collected metrics will include costs associated with initial hospitalization, surgical duration, devices utilized during the procedure, length of stay, and readmissions.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - C.H.U. of Angers, Angers
  - C.H.U. of Clermont-Ferrand, Clermont-Ferrand
  - C.H.U. of Limoges, Limoges
  - C.H.U. of Poitiers, Poitiers
  - C.H.U. Tours, Tours

REFERENCES:
- [Derived] Jayle C, Allain G, Buono A, Dang Van S, D'Ostrevy N, Kermen S, Picardo A, Pelras A, Drux J, Corbi P, Billot M, Frasca D. Reduction of the risk of complete sternotomy scar dehiscence in cardiac surgery: a protocol for a randomised, open-label multicentre clinical investigation comparing negative pressure wound therapy (NPWT) versus standard dressing (PRISTER study). BMJ Open. 2025 Nov 19;15(11):e104226. doi: 10.1136/bmjopen-2025-104226. PMID 41263903